CLINICAL TRIAL: NCT04641962
Title: A Randomized, Double-blind, Placebo-controlled Phase 2 Study to Assess the Efficacy, Safety and Tolerability of ASP0367 in Participants With Primary Mitochondrial Myopathy
Brief Title: A Study to Evaluate ASP0367 in Participants With Primary Mitochondrial Myopathy
Acronym: MOUNTAINSIDE
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Due to failure to meet the pre-specified criteria for efficacy
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0367-CL-1201
Record Dates: First submitted 2020-11-19; First posted 2020-11-24 (Actual); Results first posted 2025-06-17 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Primary Mitochondrial Myopathy
Keywords: ASP0367; fatigue; exercise intolerance; muscle weakness; Primary Mitochondrial Myopathy
MeSH Terms: conditions — Fatigue; Muscle Weakness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double blind treatment period: Participant, Caregiver, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- DBT Bocidelpar 30 mgs (Experimental): Participants received Bocidelpar 30 milligrams (mgs) orally once daily during the double blind treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
  Interventions: Drug: Bocidelpar
- DBT Bocidelpar 75mgs (Experimental): Participants received Bocidelpar 75 mg orally once daily during the DB treatment period.. The Participants were followed up for another 4 weeks after the completion of treatment period.
  Interventions: Drug: Bocidelpar
- DBT: Placebo to OLE Period: Bocidelpar 30 mg (Placebo Comparator): Participants received Bocidelpar matching placebo orally once daily during the DB treatment period and received 30 mg ASP0367 in the OLE period.
  Interventions: Drug: Bocidelpar; Drug: Placebo
- DBT Bocidelpar 30 mg or 75mg to Open label Extension Period: Bocidelpar 30 mg (Experimental): Participants received Bocidelpar 30 mg or 75 mg orally once daily during the DB treatment period and received 30 mg Bocidelpar in the OLE period.
  Interventions: Drug: Bocidelpar

INTERVENTIONS:
Drug: Bocidelpar — Oral
  Other Names: MA-0211; ASP0367
Drug: Placebo — Oral
  Arms: DBT: Placebo to OLE Period: Bocidelpar 30 mg

SUMMARY:
The purpose of this study was to evaluate the dose response of Bocidelpar on functional improvement relative to placebo, safety, and tolerability in participants with Primary Mitochondrial Myopathy.

DETAILED DESCRIPTION:
Efficacy (i.e., functional improvement) was assessed by a functional motor test, 6-minute walk test (6MWT). The study consisted of the following portions: screening (4 weeks); double-blind treatment period with 2 doses of Bocidelpar vs matching placebo (24 weeks) and follow up (4 weeks).

Participants were randomly placed into 1 of 3 arms (Bocidelpar 30 mgs, Bocidelpar 75 mgs or placebo).

ELIGIBILITY:
Inclusion Criteria:

* Participant agrees and is able to adhere to the study requirements for the length of the study, including performing 6MWT.
* Diagnosed with primary mitochondrial myopathy (PMM), consisting of the following:

  * Molecular genetic abnormality (i.e., nuclear or mitochondrial) known to be associated with mitochondrial dysfunction (such as, but not limited to, mitochondrial DNA (mtDNA) single deletions in chronic progressive external ophthalmoplegia (CPEO) and Kearns-Sayre syndrome (KSS); mtDNA m.3243 A > G pathogenic nuclear or mitochondrial genome variants demonstrated to cause primary mitochondrial disease), and
  * Participant reported symptoms (i.e., muscle weakness, fatigue and exercise intolerance) or physical examination findings of myopathy that are the predominant symptoms of the participant's mitochondrial disorder.
* Participant has been on stable dose regimen of coenzyme Q10 (CoQ10), carnitine, creatine, or other mitochondrial disease- focused vitamins or supplemental therapies for the treatment of symptoms of the mitochondrial disease for at least 3 months prior to randomization and intends to stay on a stable dose for duration of study period.
* Participant has been on stable exercise regimen within 4 weeks prior to randomization and intends to stay on a stable regimen for duration of study period (for participants who participate in a regular exercise regimen).
* Female participant is not pregnant and at least one of the following conditions apply:

  * Not a woman of childbearing potential (WOCBP).
  * WOCBP who agrees to follow the contraceptive guidance from the time of informed consent through at least 30 days after final study treatment administration.
* Female participant must agree not to breastfeed starting at screening and throughout the study period and for 30 days after final study treatment administration.
* Female participant must not donate ova starting at first dose of IP and throughout the study period and for 30 days after final study treatment administration.
* Male participant with female partner(s) of childbearing potential (including breastfeeding partner) must agree to use contraception throughout the treatment period and for 30 days after final study treatment administration.
* Male participant must not donate sperm during the treatment period and for 30 days after final study treatment administration.
* Male participant with pregnant partner(s) must agree to remain abstinent or use a condom for the duration of the pregnancy throughout the study period and for 30 days after final study treatment administration.
* Participant agrees not to participate in another interventional study while participating in the present study.

Exclusion Criteria:

* Participant has additional signs and/or symptoms due to non-myopathic process (e.g., cerebellar dysfunctions, movement disorder, peripheral neuropathy, stroke or other) or a gait problem not attributed to the myopathy that would interfere with the participant's performance during 6MWT or 5 times sit to stand (5XSTS).
* Participant has received any investigational therapy within 28 days or 5 half-lives, whichever is longer, prior to screening.
* Participant has any condition, which makes the participant unsuitable for study participation.
* Participant has cardiac troponin I (cTnI) > upper limit of normal (ULN) at screening.
* Participant has estimated glomerular filtration rate (eGFR) calculated by the chronic kidney disease epidemiology collaboration equation < 60 milliliter per minute per 1.73-meter square at screening or a history of chronic kidney disease stage 3 or greater.
* Participant has at screening*: total bilirubin (TBL) > ULN or transaminase(s) (aspartate aminotransferase [AST] or alanine aminotransferase [ALT]) > ULN in the absence of elevations in CK. Participants who have a slightly elevated TBL and/or ALT and/or AST and are suitable candidates for the study may be enrolled after discussion of the case with the medical monitor and completion of further evaluation as warranted.
* Participant has psychiatric conditions such as schizophrenia, bipolar disorder or major depressive disorder that has not been under control within 3 months prior to screening.
* Participant has a history of suicide attempt, suicidal behavior or has any suicidal ideation within 1 year prior to screening that meets criteria at a level of 4 or 5 by using the Columbia- Suicide Severity Rating Scale (C-SSRS) or who is at significant risk to commit suicide.
* Participant has severe behavioral or cognitive problems that preclude participation in the study.
* Participant has undergone an in-patient hospitalization that precludes participation in the study, within the 30 days prior to the randomization.
* Participant has a planned hospitalization or a surgical procedure during the study, which may affect the study assessments.
* Participant has clinically significant and unstable respiratory disease and/or cardiac disease (medical history or current clinical findings), or prior interventional cardiac procedure (e.g. cardiac catheterization, angioplasty/percutaneous coronary intervention, balloon valvuloplasty, etc.) within 3 months prior to randomization. Participants with pacemakers are allowed in the study per investigator's discretion and after discussion with the medical monitor, and as long as it is used for prevention and there is no underlying cardiac dysfunction.
* Participant has a corrected mean QT interval using Fridericia's correction (QTcF) > 450 msec for male participants and > 480 msec for female participants at screening or randomization. If QTcF exceeds these limits, one additional triplicate ECG can be repeated on the same day in order to determine the participant's eligibility.
* ECG evidence of acute ischemia, atrial fibrillation or active conduction system abnormalities. The following conduction system abnormalities may be permitted per the investigator's discretion, only after discussing the case with the medical monitor:

  * First degree atrioventricular (AV)- block
  * Second degree AV-block Type 1 (Mobitz Type 1/Wenckebach type)
  * Right bundle branch block
  * Left fascicular block
  * Bi-fascicular block
* Participant requires any ventilatory support, inclusive of any respiratory device to support breathing such as home ventilators and any form of non-invasive positive pressure ventilation (including continuous positive airway pressure [CPAP], bilevel positive airway pressure [BiPAP], and average volume-assured pressure support [AVAPS]). Participants who require oxygen therapy (even by low flow nasal cannula [LFNC]) are not candidates for this study.
* Participant has severe vision impairment that may interfere with their ability to complete all study requirements.
* Participant has an intractable seizure disorder that may interfere with their ability to complete all study requirements.
* Active malignancy or any other cancer from which the participant has been disease-free for < 5 years, except for curative treated localized non-melanoma skin cancer (e.g., basal cell or squamous cell carcinoma).
* Participant has a solid organ transplant and/or is currently receiving treatment with therapy for immunosuppression.
* Participant has severe scoliosis or kyphoscoliosis that significantly impair respiratory capacity and pulmonary function tests or limit positioning due to pain who would be likely to require orthopedic surgical intervention within a year after study randomization.
* Participant has a positive test for human immunodeficiency virus (HIV), hepatitis B or hepatitis C infection at screening.
* Participant has previously received Bocidelpar.
* Participant has a history of active substance abuse within 1 year prior to randomization.
* Participant has used any peroxisome proliferator-activated receptor (PPAR) ligands such as fibrates and thiazolidinediones within 4 weeks prior to randomization.
* Participant has initiated the use of CoQ10, carnitine, creatine or other mitochondrial disease-focused supplements for the treatment of symptoms of the mitochondrial disease within 3 months prior to study randomization.
* Participant has a known or suspected hypersensitivity to Bocidelpar or any components of the formulation used.
* Participant has symptomatic coronavirus disease 2019 (COVID-19) infection within 3 months prior to study randomization that required treatment (Monoclonal antibodies, ventilator support, hospitalization) and/or led to long-term sequelae or lingering symptoms.
* Participant has body mass index (BMI) below 17 kg/ m^2 or above 35 kg/ m^2 at screening.
* Participant has signs or symptoms of bulbar weakness, such as dysphagia, dysphonia, hoarseness or drooling/sialorrhea, due to either neuropathy or myopathy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2021-05-24 (Actual); Primary Completion 2024-05-08 (Actual); Study Completion 2024-05-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Senior Medical Director, Study Director — Astellas Pharma Inc
Locations (11):
- United States (11):
  - University of California, San Diego, La Jolla, California
  - Stanford University Medical Center, Stanford, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Massachusetts General Hospital, Boston, Massachusetts
  - Columbia University Irving Medical Center, New York, New York
  - Akron Children's Hospital, Akron, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Baylor College of Medicine, Houston, Texas
  - University of Texas Health Science Center at Hosuton, Houston, Texas
  - Seattle Children's Hospital, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No
Access to anonymized individual participant level data will not be provided for this trial. Further details on Astellas' data sharing policy can be found at https://www.clinicaltrials.astellas.com/transparency/.

REFERENCES:
- See also: Link to plain language summary of the study on the Trial Results Summaries website. — https://www.trialsummaries.com/Study/StudyDetails?id=14582&tenant=MT_AST_9011
- See also: Link to results and other applicable study documents on the Astellas Clinical Trials website. — https://www.clinicaltrials.astellas.com/study/0367-CL-1201

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with Primary Mitochondrial Myopathy were enrolled in the study.
Pre-assignment Details: Participants meeting all inclusion & no exclusion criteria were enrolled. Protocol version 7.0 included 4-week (wk) screening, 2 week_phase 2 dose selection portion, up to 52-wk double-blind treatment (DBT), 24-week open-label extension (OLE) & 4 wk follow-up (FU), totaling to 84 wks. Protocol v9.0: modified to 4-week screening, 24-wk DBT, 4-wk FU. Some participants received DB treatment up to 52 weeks, resulting in efficacy reported for up to 24 weeks and safety for up to 52 wks.
Groups:
- DBT: Bocidelpar 30 mg: Participants received Bocidelpar 30 mgs orally once daily during the double blind treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- DBT: Bocidelpar 75 mg: Participants received Bocidelpar 75 mg orally once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- Bocidelpar 30 mg or 75mg to Open Label Extension Period: Bocidelpar 30 mg: Participants received Bocidelpar 30 mg or 75 mg orally once daily during the DB treatment period and received 30 mg Bocidelpar in the OLE period.
- DBT: Placebo: Participants received Bocidelpar matching placebo orally once daily during the DB period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- Placebo to OLE Period: Bocidelpar 30 mg: Participants received Bocidelpar matching placebo orally once daily during the DB period and received 30mg Bocidelpar in the OLE period.
Period: DBT Period: Up to 52 Weeks
Arm/Group | DBT: Bocidelpar 30 mg | DBT: Bocidelpar 75 mg | Bocidelpar 30 mg or 75mg to Open Label Extension Period: Bocidelpar 30 mg | DBT: Placebo | Placebo to OLE Period: Bocidelpar 30 mg
Started | 12 | 11 | 0 | 11 | 0
Completed | 5 | 5 | 0 | 3 | 0
Not Completed | 7 | 6 | 0 | 8 | 0
Not completed — Miscellaneous | 5 | 3 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Not completed — Protocol deviation | 1 | 0 | 0 | 2 | 0
Not completed — Death | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 3 | 0 | 2 | 0
Period: OLE Treatment Period: Up to 76 Weeks
Arm/Group | DBT: Bocidelpar 30 mg | DBT: Bocidelpar 75 mg | Bocidelpar 30 mg or 75mg to Open Label Extension Period: Bocidelpar 30 mg | DBT: Placebo | Placebo to OLE Period: Bocidelpar 30 mg
Started | 0 | 0 | 10 | 0 | 3
Completed | 0 | 0 | 5 | 0 | 2
Not Completed | 0 | 0 | 5 | 0 | 1
Not completed — Miscellaneous | 0 | 0 | 4 | 0 | 1
Not completed — Death | 0 | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set (SAF): All randomized participants who received at least 1 dose of study drug or placebo.
Groups:
- DBT Bocidelpar 30 mg: Participants received Bocidelpar 30 mg orally once daily during the double blind treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- DBT Bocidelpar 75 mg: Participants received Bocidelpar 75 mg orally once daily during the DB period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- Total: Total of all reporting groups
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo | Total
Number analyzed (Participants) | 12 | 11 | 11 | 34
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.0 (14.2) | 33.8 (11.4) | 41.7 (12.3) | 38.2 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 8 | 7 | 21
  Male | 6 | 3 | 4 | 13
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 11 | 10 | 11 | 32
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 2 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 11 | 9 | 32
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
6 minute walk test (6MWT) [Mean (Standard Deviation); unit: Meters] — 6MWT assessed functional capacity and endurance by measuring the distance walked in 6 minutes. This test helped to assess exercise tolerance, physical fitness, disease progression, and treatment effectiveness in individuals with myopathy. The total distance walked by a participant, as well as distance per minute was calculated by rounding to the nearest meter.
  Meters | 396.3 (104.7) | 390.0 (110.6) | 422.1 (70.5) | 402.6 (95.2)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Distanced Walked During a 6 Minute Walk Test (6MWT).
Description: 6MWT assessed functional capacity and endurance by measuring the distance walked in 6 minutes. This test helped to assess exercise tolerance, physical fitness, disease progression, and treatment effectiveness in individuals with myopathy. The total distance walked by a participant, as well as distance per minute was calculated by rounding to the nearest meter.
Time Frame: Baseline, week 24
Population: Full analysis set (FAS) All randomized participants who received at least 1 dose of study drug or placebo and had at least 1 post-baseline efficacy measurement. FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Meters
Groups:
- DBT Bocidelpar 30 mg: Participants received Bocidelpar 30 mg orally once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 11 | 11 | 10
Meters | 25.3 (21.4) | 28.6 (73.3) | 17.7 (47.8)

2. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: An Adverse event (AE) was any untoward medical occurrence in a participant administered a study drug, and which dint have to have a causal relationship with this treatment. An AE could therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom or disease (new or exacerbated) temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. TEAE was defined as an AE observed after starting administration of the study drug through 28 days after the last dose.
Time Frame: From first dose up to week 52
Population: SAF
Measure: Number; unit: Participants
Groups:
- DBT Bocidelpar 75 mg: Participants received Bocidelpar 75 mg orally once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- Bocidelpar 30 or 75 mg: Participants received Bocidelpar any dose 30 or 75 mg orally once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | Bocidelpar 30 or 75 mg | DBT: Placebo
Number analyzed (Participants) | 12 | 11 | 23 | 11
Participants | 11 | 11 | 22 | 11

3. Primary Outcome: Number of Participants With Suicidal Ideation and/ or Behavior as Assessed by Columbia-Suicide Severity Rating Scale (C-SSRS)
Description: The C-SSRS was a questionnaire used for suicide risk assessment. Affirmative or negative responses were provided to items 1 to 5 for suicidal ideation (1. Wish to be dead, 2. Non-specific active suicidal thoughts, 3. Active suicidal ideation with any methods [not plan] without intent to act, 4. Active suicidal ideation with some intent to act, without specific plan, 5. Active suicidal ideation with specific plan and intent) and items 6 to 10 for suicide behavior (6. Preparatory acts or behavior, 7. Aborted attempt, 8. Interrupted attempt, 9. Actual attempt, 10. Completed suicide). The overall data was reported.
Time Frame: From the first dose up to week 52
Population: SAF
Measure: Number; unit: Participants
Groups:
- DBT Bocidelpar 75 mg: Participants received Bocidelpar 75 mg orally once daily during the DB treatment period.. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | Bocidelpar 30 or 75 mg | DBT: Placebo
Number analyzed (Participants) | 12 | 11 | 23 | 11
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Change From Baseline in Quality of Life in Neurological Disorders (Neuro-QoL) Short Form Fatigue Score
Description: The Neuro-QoL Short Form Fatigue score was an 8-item self- assessment questionnaire evaluating the perception of fatigue and its impact in daily life activities. Participants had five response options for each item: 1=Never, 2=Rarely, 3=Sometimes, 4=Often, 5=Always. The questionnaire was scored by adding the response to each of the item and then transformed into T-scores based on the scoring manual with a score range of minimum=29.5, maximum=74.1. T-score distributions rescaled raw scores into standardized scores with a mean of 50 and a SD of 10. Higher scores indicated a greater level of fatigue.
Time Frame: Baseline, week 24
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: T score
Groups:
- DBT: Bocidelpar 30 mg: Participants received Bocidelpar 30 mg orally once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT: Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 8 | 8 | 6
T score | -4.04 (4.59) | -1.09 (4.40) | -2.82 (8.63)

5. Secondary Outcome: Change From Baseline in Neuro-QoL Short Form Lower Extremity Function (Mobility) Scores
Description: The Neuro-QoL Short Form Lower Extremity Function (Mobility) score was an 8-item self- assessment questionnaire evaluating the functioning of one's lower extremities. Participants responded to questions on a 1-5 scale. Participants had five response options for each item: 1=Unable to do,2=With much difficulty,3=With some difficulty,4=With a little difficulty, 5=Without any difficult. The questionnaire was scored by adding the response to each of the item and then transformed into T-scores based on the scoring manual with a score range of minimum=16.5, maximum=58.6. T-score distributions rescaled raw scores into standardized scores with a mean of 50 and a SD of 10. Higher scores indicated better function.
Time Frame: Baseline, week 24
Population: FAS with available data were analyzed.
Measure: Mean (Standard Deviation); unit: T scoree
Groups:
- DBT Bocidelpar 30 mg: Participants received Bocidelpar 30 mg orally once daily during the DB period. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 8 | 8 | 6
T scoree | 2.49 (3.36) | 1.68 (3.67) | 2.50 (6.02)

6. Secondary Outcome: Change From Baseline in Time to Perform the 5 Times Sit to Stand (5XSTS) Test
Description: The 5XSTS test was a functional assessment that measured the time taken to stand up from a seated position five times in a row, as quickly as possible. The duration from the time instructor indicated "Go" until the time participant's body touched the chair following the fifth repetition was recorded and reported.
Time Frame: Baseline, week 24
Population: FAS with available participants were analyzed.
Measure: Mean (Standard Deviation); unit: Seconds
Groups:
- DBT Bocidelpar 30 mg: Participants received DBT Bocidelpar 30 mg orally once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 8 | 7 | 6
Seconds | -1.1 (2.6) | -0.9 (2.6) | -1.5 (2.7)

7. Secondary Outcome: Number of Participants With Patient's Global Impression of Change (PGIC) Score at Week 24
Description: The PGIC scale evaluated the participant's symptom and assessed if there had been any improvement or decline in clinical status. The participant rated their perceived change on a 7-point scale, with 1 indicating very much improved, 2 = Much Improved, 3=Minimally Improved, 4= No Change, 5=Minimally Worse, 6=Much Worse and 7 indicating 'very much worse".
Time Frame: Week 24
Population: FAS with available data were analyzed.
Measure: Number; unit: participants
Groups:
- DBT Bocidelpar 30 mg: Participants received Bocidelpar 30 mg orally once daily during the DB treatment period.. The Participants were followed up for another 4 weeks after the completion of treatment period.
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 9 | 8 | 7
participants
  Very Much Improved | 1 | 0 | 0
  Much Improved | 1 | 1 | 2
  Minimally Improved | 3 | 2 | 3
  No Change | 4 | 4 | 1
  Minimally Worse | 0 | 1 | 1
  Much Worse | 0 | 0 | 0
  Very Much Worse | 0 | 0 | 0

8. Secondary Outcome: Number of Participants With Change From Baseline in Patient Global Impression of Severity (PGIS) at Week 24
Description: PGIS score was a patient-reported measure that reflected the individual's overall perception of the severity of their condition on a Likert scale. PGIS score were calculated as -1= mild change from baseline, -2=moderate change from baseline,-3=severe change from baseline,0= none, 1= mild, 2= moderate and 3= severe. The questionnaire asked the participant to best describe the severity of the participant's most bothersome pre-defined symptom over the past week.
Time Frame: Baseline, week 24
Population: FAS with available data were analyzed.
Measure: Number; unit: Participants
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 8 | 8 | 6
Participants
  -3 | 0 | 0 | 0
  -2 | 1 | 0 | 0
  -1 | 3 | 3 | 4
  0 | 4 | 5 | 2
  1 | 0 | 0 | 0
  2 | 0 | 0 | 0
  3 | 0 | 0 | 0

9. Secondary Outcome: Change From Baseline in Modified Fatigue Impact Scale (MFIS)
Description: MFIS was a self-reported questionnaire designed to evaluate the impact of fatigue on physical, cognitive and psychosocial functioning. The MFIS consisted of 21 items scored 0-4 (0=Never, 1=Rarely, 2=Sometimes, 3=Often, and 4=Almost always). The total MFIS score ranged from 0 to 84, with three subscales: Physical range 0-36, Cognitive range 0-40, and Psychosocial range 0-8. Higher scores indicated higher level of fatigue.
Time Frame: Baseline, week 24
Population: FAS with available data was analyzed.
Measure: Mean (Standard Deviation); unit: Score on a Scale
Arm/Group | DBT Bocidelpar 30 mg | DBT Bocidelpar 75 mg | DBT: Placebo
Number analyzed (Participants) | 8 | 8 | 6
Score on a Scale
  Physical | -3.4 (3.2) | -1.4 (5.0) | -4.8 (4.9)
  Cognitive | -1.9 (6.7) | 0.0 (7.8) | -0.7 (4.0)
  Psychosocial | -0.8 (1.7) | -0.6 (1.1) | -1.8 (2.1)
  Total Score | -6.0 (8.0) | -2.0 (11.7) | -7.3 (9.8)

ADVERSE EVENTS:
Time Frame: Serious/Non Serious AE: From first dose up to week 76 All cause mortality: From randomization up to 76 weeks.
Description: AE occurring after administration of study drug up to 28 days after last dose based on protocol version under which participants were enrolled. • Protocol Version 7.0: Included 52-week DBT period, 24-week OLE & 4-week follow-up period. • Protocol Version 9.0: Included 24-week DBT period & 4-week follow-up period. Data on AE was collected up to 76 weeks. The timing of last dose varied among participants, as a result, some participants remained in study for longer than 24 weeks.
Groups:
- DBT Placebo: Participants received Bocidelpar matching placebo orally once daily during the DB period. The Participants were followed up for another4 weeks after the completion of treatment period.
- DBT Bocidelpar 75 mg: Participants received Bocidelpar 75 mg once daily during the DB treatment period. The Participants were followed up for another 4 weeks after the completion of treatment period.
- Placebo to Open-label Extension Period: Bocidelpar 30 mg: Participants received Bocidelpar matching placebo orally once daily during the DB treatment period and received 30 mg Bocidelpar in the OLE period.
- Bocidelpar 30 mg or 75 mg to Open-label Extension Period: Bocidelpar 30 mg: Participants received Bocidelpar 30 mg or 75 mg orally once daily during the DB treatment period and received 30 mg Bocidelpar in the OLE period.
Arm/Group | DBT Placebo | DBT: Bocidelpar 30 mg | DBT Bocidelpar 75 mg | Placebo to Open-label Extension Period: Bocidelpar 30 mg | Bocidelpar 30 mg or 75 mg to Open-label Extension Period: Bocidelpar 30 mg
All-Cause Mortality (participants affected / at risk) | 0/11 | 1/12 | 0/11 | 0/3 | 1/10
Serious Adverse Events (participants affected / at risk) | 1/11 | 1/12 | 2/11 | 0/3 | 1/10
Other Adverse Events (participants affected / at risk) | 11/11 | 11/12 | 11/11 | 3/3 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBT Placebo (N=11) | DBT: Bocidelpar 30 mg (N=12) | DBT Bocidelpar 75 mg (N=11) | Placebo to Open-label Extension Period: Bocidelpar 30 mg (N=3) | Bocidelpar 30 mg or 75 mg to Open-label Extension Period: Bocidelpar 30 mg (N=10)
Arrhythmia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
MELAS syndrome (Congenital, familial and genetic disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Troponin I increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | DBT Placebo (N=11) | DBT: Bocidelpar 30 mg (N=12) | DBT Bocidelpar 75 mg (N=11) | Placebo to Open-label Extension Period: Bocidelpar 30 mg (N=3) | Bocidelpar 30 mg or 75 mg to Open-label Extension Period: Bocidelpar 30 mg (N=10)
Bundle branch block (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MELAS syndrome (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Progressive external ophthalmoplegia (Congenital, familial and genetic disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Asthenopia (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Astigmatism (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Choroidal neovascularisation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diplopia (Eye disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Eye movement disorder (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Strabismus (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aphthous ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 3 (3) | 0 (0) | 3 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Epigastric discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Food poisoning (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 0 (0)
Salivary hypersecretion (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Toothache (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Asthenia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Feeling cold (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Influenza like illness (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Vessel puncture site bruise (General disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (4) | 2 (2) | 4 (4) | 0 (0) | 6 (6)
Conjunctivitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal viral infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymph gland infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pharyngitis streptococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Viral infection (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Immunisation reaction (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Ligament sprain (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1)
Lip injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Post vaccination fever (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Procedural nausea (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular access site bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vascular access site pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 3 (4) | 1 (1) | 0 (0) | 3 (4)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 2 (3)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 3 (4) | 2 (3) | 0 (0) | 3 (5)
Blood phosphorus decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood triglycerides increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glutamate dehydrogenase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Grip strength decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lipase increased (Investigations) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transaminases increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Troponin T increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyslipidaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Mastication disorder (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Tendon pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Balance disorder (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disturbance in attention (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 3 (5) | 0 (0) | 0 (0) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Sleep disorder (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dysuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urine odour abnormal (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Amenorrhoea (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Vulvovaginal burning sensation (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Snoring (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Hot flush (Vascular disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pallor (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
The study was terminated due to futility after protocol version 9.0 was introduced. Some participants received treatment for up to 52 weeks, resulting in efficacy reported for up to 24 weeks and safety for up to 52 weeks.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Institute and/or Principal Investigator may publish trial data generated at their specific study site after Sponsor publication of the multi-center data. Sponsor must receive a site's manuscript prior to publication for review and comment as specified in the Investigator Agreement.

DOCUMENTS (2):
  • Study Protocol (2024-01-24): https://cdn.clinicaltrials.gov/large-docs/62/NCT04641962/Prot_000.pdf
  • Statistical Analysis Plan (2024-07-09): https://cdn.clinicaltrials.gov/large-docs/62/NCT04641962/SAP_001.pdf